CLINICAL TRIAL: NCT03438747
Title: An Assessment of P-15L Bone Graft in Transforaminal Lumbar Interbody Fusion With Instrumentation
Brief Title: P-15L Bone Graft in Transforaminal Lumbar Interbody Fusion With Instrumentation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CeraPedics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CP-1006; NCT03502057 (obsolete NCT alias)
Record Dates: First submitted 2018-02-13; First posted 2018-02-20 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- P-15L Bone Graft (Experimental): The investigational group will be treated with P-15L Bone Graft in an instrumented TLIF
  Interventions: Device: P-15L Bone Graft
- Local autologous bone (Active Comparator): The active control group will be treated with local autologous bone in an instrumented TLIF
  Interventions: Other: Local autologous bone in a TLIF with Instrumentation

INTERVENTIONS:
Device: P-15L Bone Graft — The investigational group will be treated with P-15L in an instrumented TLIF
  Arms: P-15L Bone Graft
Other: Local autologous bone in a TLIF with Instrumentation — The active control group will be treated local autologous bone in an instrumented TLIF
  Arms: Local autologous bone

SUMMARY:
The aim of this trial is to evaluate if P-15L bone graft (investigational device) is not inferior in effectiveness and safety to local autologous bone (and allograft where necessary) as an extender (control device) when applied in instrumented transforaminal lumbar interbody fusion (TLIF) in subjects with degenerative disc disease (DDD). In addition to the general overall objective, a sub-group analysis will be performed on the high-risk subject population (tobacco use, obesity, diabetes), as previous studies have shown negative effects of smoking, obesity and diabetes on fusion and bone healing, increased peri/postoperative complications, and lower patient-reported outcome scores.

ELIGIBILITY:
Inclusion Criteria (abbreviated):

Skeletally mature adults between 22 and 80 years old (inclusive);

Back pain with radicular symptoms as evidenced by leg pain, confirmed by history and physical exam;

Oswestry Low Back Pain Disability Questionnaire score of ≥ 35;

Involved disc(s) between L2 and S1;

Exclusion Criteria (abbreviated):

Significant metabolic disease that in the surgeon's opinion might compromise bone growth such as osteoporosis, osteopenia, or osteomalacia;

Active malignancy;

Nondiscogenic source of symptoms (e.g. tumor, etc.);

Multiple level symptomatic degenerative disc disease where more than one level requires fusion;

Previous spinal instrumentation or a previous interbody fusion procedure at the involved level;

More than one level to be fused

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Secondary surgical intervention | 72 Months
  No index level secondary surgical intervention
Fusion | 72 Months
  Achievement of fusion (Fusion is defined as evidence of bridging trabecular bone between the vertebral bodies by CT scan)
Oswestry Disability Index (ODI) | 72 Months
  At least 15-point improvement in Oswestry Disability Index (ODI)
Neurological deficit | 72 Months
  No new or worsening, persistent neurological deficit
No serious device-related adverse event | 72 Months
  No serious device-related adverse event

SECONDARY OUTCOMES:
Time to Fusion | 24 months
  The distribution of visits (month 6, 12, or 24) at which fusion is confirmed is the same for the investigational and control devices.
VAS pain scores | 72 months
  Pain at back and pain at legs will be measured by a 100-point Visual Analog Scale (VAS)
Physical Function and Mental Health Composite Scores | 72 months
  SF-12 and changes over time

CONTACTS AND LOCATIONS:
Locations (34):
- United States (34):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Glendale Adventist Medical Center, Glendale, California
  - Keck School of Medicine USC, Los Angeles, California
  - UC Irvine Medical Center, Orange, California
  - UC Davis Spine Center, Sacramento, California
  - Cedars-Sinai, West Hollywood, California
  - Center for Spine and Orthopedics, Thornton, Colorado
  - UConn Health, Farmington, Connecticut
  - St. Francis Hospital and Medical Center, Hartford, Connecticut
  - University of South Florida, Tampa, Florida
  - Florida Orthopaedic Institute, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Indiana Spine Group, Carmel, Indiana
  - OrthoIndy, Indianapolis, Indiana
  - Norton Leatherman Spine Center, Louisville, Kentucky
  - Orthopaedic Institute of Western Kentucky, Paducah, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - University Of Buffalo, Buffalo, New York
  - The Orthopedic Center at Mount Sinai West, New York, New York
  - SUNY Upstate Medical Center, Syracuse, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Rothman Institute, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Canter, Pittsburgh, Pennsylvania
  - Austin Neurosurgeons, Austin, Texas
  - Texas Back Institute, Plano, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - Swedish Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Harrop JS, O'Toole JE, Steinmetz MP, Sasso RC, Chaput CD, Strenge KB, Maislin G, Mullin JP, Freeman TB, Guanciale A, Lantner H, Janssen ME, Schwartz DG, Small JM, Hsu WK, Arnold PM. P-15 Peptide Enhanced Bone Graft in Transforaminal Lumbar Interbody Fusion: A Randomized, Controlled, Investigational Device Exemption Study Demonstrating Improved Composite Clinical Success. Spine (Phila Pa 1976). 2026 Feb 15;51(4):238-247. doi: 10.1097/BRS.0000000000005579. Epub 2025 Dec 19. PMID 41307132
- [Derived] Harrop JS, Steinmetz MP, O'Toole JE, Chaput CD, Sasso RC, Strenge KB, Maislin G, Mullin JP, Freeman TB, Guanciale A, Lantner H, Janssen ME, Schwartz DG, Small JM, Hsu WK, Arnold PM. P-15 Peptide Enhanced Bone Graft Improves Time to Fusion in Transforaminal Lumbar Interbody Fusion: A Randomized, Controlled, Investigational Device Exemption Study. Spine (Phila Pa 1976). 2026 Feb 15;51(4):229-237. doi: 10.1097/BRS.0000000000005580. Epub 2025 Dec 19. PMID 41307110